CLINICAL TRIAL: NCT01957657
Title: Pharmacokinetics, Safety and Tolerability of the Combination of BI 207127 and Faldaprevir in Patients With Different Degrees of Renal Impairment in Comparison to Subjects With Normal Renal Function in a Single Center, Open-label, Parallel-group, Phase I Trial
Brief Title: Pharmacokinetics, Safety and Tolerability of the Combination of BI 207127 and Faldaprevir in Renal Impaired Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1241.32; 2013-001075-21 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-10-01; First posted 2013-10-08 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — deleobuvir; faldaprevir

ARMS (4):
- Healthy volunteers group 1 (Experimental): Healthy volunteers with normal renal function
  Interventions: Drug: BI 207127; Drug: faldaprevir
- Renal function group 2 (Experimental): Patients with mild renal impairment
  Interventions: Drug: BI 207127; Drug: faldaprevir
- Renal function group 3 (Experimental): Patients with moderate renal impairment
  Interventions: Drug: BI 207127; Drug: faldaprevir
- Renal function group 4 (Experimental): Patients with severe renal impairment
  Interventions: Drug: BI 207127; Drug: faldaprevir

INTERVENTIONS:
Drug: BI 207127 — oral administration
  Arms: Renal function group 2
Drug: faldaprevir — oral administration
  Arms: Renal function group 2
Drug: BI 207127 — oral administration
  Arms: Renal function group 4
Drug: BI 207127 — oral administration
  Arms: Healthy volunteers group 1
Drug: BI 207127 — oral administration
  Arms: Renal function group 3
Drug: faldaprevir — oral administration
  Arms: Renal function group 3
Drug: faldaprevir — oral administration
  Arms: Healthy volunteers group 1
Drug: faldaprevir — oral administration
  Arms: Renal function group 4

SUMMARY:
The objective of the trial is to investigate the effect of different degrees of renal impairment on the pharmacokinetics and safety of the combination of BI 207127 and faldaprevir after 3 days of dosing (BI 207127 bid, faldaprevir qd) and a single dose of BI 207127 and faldaprevir on day 4.

ELIGIBILITY:
Inclusion criteria:

* Healthy volunteers (males and females) or patients with impaired renal function (estimated glomerular filtration rate (eGFR) between 89 and 15) in relatively good health as determined by past medical history, physical examination, vital signs, ECG and laboratory assessments (aside from abnormalities specific for renal impairment)
* Age from 18 to 79 years
* Subjects must be able to understand and comply with study requirements

Exclusion criteria:

* Any relevant deviation from healthy conditions for healthy volunteers
* Subjects with significant diseases other than renal impairment will be excluded. A significant disease is defined as a disease which in the opinion of the investigator:

  * put the patient at risk because of participation in the study
  * may influence the results of the study
  * may influence the patients ability to participate in the study
  * is not in a stable condition
* Diabetic or hypertensive patients can be entered in this trial if the disease is not significant according to these criteria

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1241.32.1 Boehringer Ingelheim Investigational Site, Kiel, Germany

REFERENCES:
- [Derived] Huang F, Moschetti V, Lang B, Halabi A, Petersen-Sylla M, Yong CL, Elgadi M. Pharmacokinetics, safety, and tolerability of faldaprevir in patients with renal impairment. Antimicrob Agents Chemother. 2015 Jan;59(1):251-7. doi: 10.1128/AAC.03359-14. Epub 2014 Oct 27. PMID 25348520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patient groups with renal impairment were to be investigated consecutively starting with the mildly impaired, followed by the moderately impaired, and the severely impaired group. Normal renal function patients were to be investigated last. The trial was terminated after four patients were enrolled and completed.
Groups:
- Deleobuvir + Faldaprevir, Mild Renal Impairment: Multiple doses of deleobuvir, immediate release tablet, plus faldaprevir, soft gelatin capsule, were planned to be administered over 4 days to patients with mild renal impairment.
  Administration of 600 mg deleobuvir bid and 120 mg faldaprevir, qd on Days 1 to 3 (with a single loading dose of 240 mg faldaprevir qd on Day 1) and 600 mg deleobuvir qd and faldaprevir 120 mg qd on Day 4.
  All four patients had mild renal impairment, i.e., estimated glomerular filtration rate (eGFR) of 60-89 mL/min.
Period: Overall Study
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated Set, (TS) included all enrolled subjects, who had taken at least one dose of trial medication.
Groups:
- Deleobuvir + Faldaprevir, Mild Renal Impairment: Multiple doses of deleobuvir plus faldaprevir were planned to be administered over 4 days to patients with mild renal impairment.
  Administration of 600 mg deleobuvir bid and 120 mg faldaprevir qd on Days 1 to 3 (with a single loading dose of 240 mg faldaprevir qd on Day 1) and 600 mg deleobuvir qd and faldaprevir 120 mg qd on Day 4.
  All four patients had mild renal impairment, i.e., estimated glomerular filtration rate (eGFR) of 60-89 mL/min.
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  Germany | 4

OUTCOME MEASURES:

1. Primary Outcome: AUC 0-infinity (Area Under the Concentration-time Curve of Deleobuvir (BI 207127) in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: Blood sampling for Pharmacokinetic (PK) profiles was performed after the last dosing of the combination treatment on Day 4 at the following time points: for deleobuvir (BI 207127) and metabolites at 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 10, 12, 24, 48 and 72 h after dosing; for faldaprevir at 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120 and 144 h after drug administration in the morning.
Time Frame: Day 4
Population: Boehringer Ingelheim decided to stop the further development of the interferon-free combination therapy for Hepatitis C and terminated the trial prematurely on 27 Dec 2013. Since the sample size achieved at trial termination was much smaller than the planned sample size the pharmacokinetic endpoints were not determined.
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 0

2. Primary Outcome: Cmax (Maximum Measured Concentration of Deleobuvir (BI 207127) in Plasma)
Description: Blood sampling for PK profiles was performed after the last dosing of the combination treatment on Day 4 at the following time points: for deleobuvir (BI 207127) and metabolites at 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 10, 12, 24, 48 and 72 h after dosing; for faldaprevir at 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120 and 144 h after drug administration in the morning.
Time Frame: Day 4
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 0

3. Secondary Outcome: Number (%) of Subjects With Drug-related Adverse Events
Description: Number (percentage) of subjects with drug-related adverse events
Time Frame: From the first drug administration until last drug administration, up to 10 days
Population: Treated set (TS) included all enrolled subjects, who had taken at least one dose of trial medication.
Measure: Number; unit: percentage of participants
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 4
percentage of participants | 25

4. Secondary Outcome: AUC 0-infinity (Area Under the Concentration-time Curve of Deleobuvir (BI 207127) Metabolite (CD 6168) in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: as for outcome 2
Time Frame: Day 4
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 0

5. Secondary Outcome: AUC 0-infinity (Area Under the Concentration-time Curve of Deleobuvir (BI 207127) Metabolite (BI 208333) in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: as for outcome 2
Time Frame: Day 4
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 0

6. Secondary Outcome: AUC 0-infinity (Area Under the Concentration-time Curve of Deleobuvir (BI 207127) Metabolite (CD 6168 Acylglucuronide) in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: as for outcome 2
Time Frame: Day 4
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 0

7. Secondary Outcome: AUC 0-infinity (Area Under the Concentration-time Curve of Faldaprevir in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: as for outcome 2
Time Frame: Day 4
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 0

8. Secondary Outcome: Cmax (Maximum Measured Concentration of Deleobuvir (BI 207127) Metabolite (CD 6168) in Plasma)
Description: as for outcome 2
Time Frame: Day 4
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 0

9. Secondary Outcome: Cmax (Maximum Measured Concentration of Deleobuvir (BI 207127) Metabolite (BI 208333) in Plasma)
Description: as for outcome 2
Time Frame: Day 4
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 0

10. Secondary Outcome: Cmax (Maximum Measured Concentration of Deleobuvir (BI 207127) Metabolite (CD 6168 Acylglucuronide) in Plasma)
Description: as for outcome 2
Time Frame: Day 4
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 0

11. Secondary Outcome: Cmax (Maximum Measured Concentration of Faldaprevir in Plasma)
Description: as for outcome 2
Time Frame: Day 4
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first drug administration until day after end of trial examination, up to 18 days
Arm/Group | Deleobuvir + Faldaprevir, Mild Renal Impairment
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deleobuvir + Faldaprevir, Mild Renal Impairment (N=4)
Nausea (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
The sponsor decided to stop the development of Hepatitis C treatments and terminated the trial prematurely on 27 Dec 2013. Due to the small sample size the pharmacokinetic endpoints were not determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.